CLINICAL TRIAL: NCT02133716
Title: Efficacy of Breast Milk Expressed Versus Sucrose Relief Procedural Pain of Venipuncture in Preterm.
Brief Title: Efficacy of Breast Milk Expressed and Sucrose in Procedural Pain in Preterm
Acronym: LACTEET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Laura Collados Gómez, Laura Collados Gómez, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LACTEET
Record Dates: First submitted 2014-04-17; First posted 2014-05-08 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2014-05

CONDITIONS: Pain; Premature Infant; Human Milk; Breastfeeding
Keywords: pain; premature infant; sucrose; breastfeeding; expressed breast milk; PIPP
MeSH Terms: conditions — Pain; Premature Birth; Breast Feeding | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- expressed breast milk (Experimental): A single dose of expressed breast milk was administered through a sterile syringe in the mouth 2 minutes before venopuncture to neonates, accompanied at all times provided the technique allows it to non-nutritive sucking and containment.
  The doses administered: 0.1ml in infants less than 27 weeks , 0.25 ml for infants 27-31 weeks , 0.5 ml for infants 32-37 weeks.
  Interventions: Other: expressed breast milk
- sucrose 24% oral (Active Comparator): A single dose of sucrose was administered through a sterile syringe in the mouth 2 minutes before venopuncture to neonates, accompanied at all times provided the technique allows it to non-nutritive sucking and containment.
  The doses administered: 0.1ml in infants less than 27 weeks , 0.25 ml for infants 27-31 weeks , 0.5 ml for infants 32-37 weeks.
  Interventions: Behavioral: sucrose 24% oral

INTERVENTIONS:
Other: expressed breast milk — The administration will be by direct instillation feeding syringe (maximum capacity 1ml) in the front of the mouth of the infant and accompanied throughout the administration of non-nutritive sucking (pacifier) and manual containing both sucrose treatment oral, as in the oral expressed breastmilk.
  A single dose prior to venipuncture of expressed breast milk given two minutes in the sequence and then will proceed to the venipuncture care nurse responsible for the child, accompanied at all times provided the technical permitted with non-nutritive sucking and containment.
  Arms: expressed breast milk
Behavioral: sucrose 24% oral — The administration will be by direct instillation feeding syringe (maximum capacity 1ml) in the front of the mouth of the infant and accompanied throughout the administration of non-nutritive sucking (pacifier) and manual containing both sucrose treatment oral, as in the oral expressed breastmilk.
  A single dose prior to venipuncture of oral sucrose 24% given two minutes in the sequence and then will proceed to the venipuncture care nurse responsible for the child, accompanied at all times provided the technical permitted with non-nutritive sucking and containment.
  Arms: sucrose 24% oral

SUMMARY:
The aim of this study is to assess the non-inferiority of non- pharmacological breast milk expressed versus oral sucrose in relief procedural pain of venipuncture in preterm neonates.

This is an experimental comparative study of non-inferiority randomized crossover, to be performed in Neonatal units of hospitals in the Community of Madrid.

The 54 pair of preterm that after the selection criteria are included in the study, they performed the randomization of the sequence and breast milk expressed receive oral or 24% sucrose.

The doses administered are: 0.1ml preterm less than 27 weeks corrected gestational age (CGA), 0.25 ml for infants 27 to 31 weeks CGA and 0.5 ml for infants of 32-37 weeks. Both groups will be accompanied by non-nutritive sucking and swaddling and administered two minutes prior to venipuncture.

The outcome variable, pain, will be determined by the scale Premature Infant Pain Profile (PIPP) and by percent of cry.

Data for the primary objective was analysed per intention to treat. This study was approved by local ethical committee.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates.
* Weight less than 2500 grams.
* Feed breastfeeding (exclusive or not) or can obtain weight expressed breastmilk .
* Be informed and consent to the parents of those infants previously requested.

Exclusion Criteria:

* Maternal use of opioids or insulin-depent
* infants with invasive artificial respiration
* infants with major congenital anomalies
* infants with grade II or IV intraventricular hemorrhage or strokes
* receiving parental sedatives or vasoactive drugs
* infants with necrotizing enterocolitis
* with surgical interventions
* infants in absolute diet
* infants with abstinence syndrome

Ages: 25 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pain neonatal | Midpoint analysis will be conducted when half the patients are recruited, at an estimated time of 12 months
  The pain neonatal will be determined by the scale Premature Infant Pain Profile (PIPP). The PIPP scale is a multidimensional measure developed to assess pain in preterm and term infants.
  It consists of three behavioral indicators (facial actions: philtrum, frowning, clenched eyes), two physiological indicators (heart rate and oxygen saturation) and two measures of development (gestational age and behavioral state). Each pointer may take four values on a scale from 0 to 3, which is subsequently added to an overall score. The score range from 0 (no pain or the presence of minimal pain) to 21 (maximum pain) in preterm.
  PIPP score was evaluated at 30 seconds after venopuncture Both the validity and reliability of this scale have been studied and proven in various studies.
  The PIPP scale will it be monitored by skilled and experienced nurses in neonatal care.

SECONDARY OUTCOMES:
Percentage of crying | Midpoint analysis will be conducted when half the patients are recruited, at an estimated time of 12 months
  Relationship between duration procedure venipuncture and the time or duration of crying(from beginning to cry until terminated.)

OTHER OUTCOMES:
Number of attempts | Midpoint analysis will be conducted when half the patients are recruited, at an estimated time of 12 months.
  Number of attempts during the venopuncture

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital University Gregorio Marañon, Madrid, Madrid, Spain

REFERENCES:
- [Background] American Academy of Pediatrics Committee on Fetus and Newborn; American Academy of Pediatrics Section on Surgery; Canadian Paediatric Society Fetus and Newborn Committee; Batton DG, Barrington KJ, Wallman C. Prevention and management of pain in the neonate: an update. Pediatrics. 2006 Nov;118(5):2231-41. doi: 10.1542/peds.2006-2277. PMID 17079598
- [Background] Bouza H. The impact of pain in the immature brain. J Matern Fetal Neonatal Med. 2009 Sep;22(9):722-32. doi: 10.3109/14767050902926962. PMID 19526425
- [Background] Bueno M, Stevens B, de Camargo PP, Toma E, Krebs VL, Kimura AF. Breast milk and glucose for pain relief in preterm infants: a noninferiority randomized controlled trial. Pediatrics. 2012 Apr;129(4):664-70. doi: 10.1542/peds.2011-2024. Epub 2012 Mar 5. PMID 22392169
- [Background] Carbajal R, Rousset A, Danan C, Coquery S, Nolent P, Ducrocq S, Saizou C, Lapillonne A, Granier M, Durand P, Lenclen R, Coursol A, Hubert P, de Saint Blanquat L, Boelle PY, Annequin D, Cimerman P, Anand KJ, Breart G. Epidemiology and treatment of painful procedures in neonates in intensive care units. JAMA. 2008 Jul 2;300(1):60-70. doi: 10.1001/jama.300.1.60. PMID 18594041
- [Background] Vinall J, Grunau RE. Impact of repeated procedural pain-related stress in infants born very preterm. Pediatr Res. 2014 May;75(5):584-7. doi: 10.1038/pr.2014.16. Epub 2014 Feb 5. PMID 24500615
- [Background] Johnston CC, Filion F, Snider L, Majnemer A, Limperopoulos C, Walker CD, Veilleux A, Pelausa E, Cake H, Stone S, Sherrard A, Boyer K. Routine sucrose analgesia during the first week of life in neonates younger than 31 weeks' postconceptional age. Pediatrics. 2002 Sep;110(3):523-8. doi: 10.1542/peds.110.3.523. PMID 12205254
- [Background] Lopez Maestro M, Melgar Bonis A, de la Cruz-Bertolo J, Perapoch Lopez J, Mosqueda Pena R, Pallas Alonso C. [Developmental centered care. Situation in Spanish neonatal units]. An Pediatr (Barc). 2014 Oct;81(4):232-40. doi: 10.1016/j.anpedi.2013.10.043. Epub 2013 Dec 2. Spanish. PMID 24290892
- [Background] Marin Gabriel MA, del Rey Hurtado de Mendoza B, Jimenez Figueroa L, Medina V, Iglesias Fernandez B, Vazquez Rodriguez M, Escudero Huedo V, Medina Malagon L. Analgesia with breastfeeding in addition to skin-to-skin contact during heel prick. Arch Dis Child Fetal Neonatal Ed. 2013 Nov;98(6):F499-503. doi: 10.1136/archdischild-2012-302921. Epub 2013 Jul 9. PMID 23839984
- [Background] Ors R, Ozek E, Baysoy G, Cebeci D, Bilgen H, Turkuner M, Basaran M. Comparison of sucrose and human milk on pain response in newborns. Eur J Pediatr. 1999 Jan;158(1):63-6. doi: 10.1007/s004310051011. PMID 9950311
- [Background] Ozdogan T, Akman I, Cebeci D, Bilgen H, Ozek E. Comparison of two doses of breast milk and sucrose during neonatal heel prick. Pediatr Int. 2010 Apr;52(2):175-9. doi: 10.1111/j.1442-200X.2009.02921.x. Epub 2009 Jul 16. PMID 19627552
- [Background] Ou-Yang MC, Chen IL, Chen CC, Chung MY, Chen FS, Huang HC. Expressed breast milk for procedural pain in preterm neonates: a randomized, double-blind, placebo-controlled trial. Acta Paediatr. 2013 Jan;102(1):15-21. doi: 10.1111/apa.12045. Epub 2012 Nov 1. PMID 23057434
- [Background] Shah PS, Herbozo C, Aliwalas LL, Shah VS. Breastfeeding or breast milk for procedural pain in neonates. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD004950. doi: 10.1002/14651858.CD004950.pub3. PMID 23235618
- [Background] Pillai Riddell RR, Racine NM, Turcotte K, Uman LS, Horton RE, Din Osmun L, Ahola Kohut S, Hillgrove Stuart J, Stevens B, Gerwitz-Stern A. Non-pharmacological management of infant and young child procedural pain. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD006275. doi: 10.1002/14651858.CD006275.pub2. PMID 21975752
- [Background] Simonse E, Mulder PG, van Beek RH. Analgesic effect of breast milk versus sucrose for analgesia during heel lance in late preterm infants. Pediatrics. 2012 Apr;129(4):657-63. doi: 10.1542/peds.2011-2173. Epub 2012 Mar 5. PMID 22392168
- [Background] Stevens B, Johnston C, Petryshen P, Taddio A. Premature Infant Pain Profile: development and initial validation. Clin J Pain. 1996 Mar;12(1):13-22. doi: 10.1097/00002508-199603000-00004. PMID 8722730
- [Background] Stevens B, Yamada J, Lee GY, Ohlsson A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD001069. doi: 10.1002/14651858.CD001069.pub4. PMID 23440783